CLINICAL TRIAL: NCT03678298
Title: Italian Register for the Study of Complicated Intra-Abdominal Infections (IRCA) Study
Brief Title: Italian Register for the Study of Complicated Intra-Abdominal Infections
Acronym: IRCA
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: World Society of Emergency Surgery (Other)
Responsible Party: Principal Investigator, Massimo Sartelli, Medical Doctor, World Society of Emergency Surgery
Other Study IDs: 1/2018
Record Dates: First submitted 2018-09-17; First posted 2018-09-19 (Actual); Last update posted 2018-09-19 (Actual); Status verified 2018-08

CONDITIONS: Complicated Intra-abdominal Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples Without DNA — Microbiological samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Epidemiological/treatment profiles — All consecutively hospitalized adult patients (older than 18 years of age) undergoing surgery, interventional drainage or conservative treatment, with diagnosis of cIAIs (defined as abdominal infections originating in an organ cavity, extending into the peritoneal space, and forming an abscess or peritonitis, will be included in the study.

SUMMARY:
The study will identify the epidemiological and treatment profiles of acute peritonitis in Italy

DETAILED DESCRIPTION:
The primary objectives of the study are: (1) the identification of specific risk factors for in-hospital mortality, in order to perfect the clinical management of patients with complicated intra-abdominal infections (cIAIs); (2) the identification of specific risk factors for multi-drug resistant organisms (MDROs) isolation in patients with cIAIs, in order to improve the adequacy of empirical antimicrobial therapy.

The secondary objectives are: (1) the description of the clinical, diagnostic and treatment profiles of patients with cIAIs in Italian surgical departments; (2) the analysis of epidemiology and patterns of antimicrobial susceptibility of the microorganisms isolated in samples in intra-operative samples of peritoneal fluid or purulent exudate/discrete abscesses in patients with cIAIs; (3) the identification of specific risk factors for post-operative complications in patients with cIAIs.

ELIGIBILITY:
Inclusion Criteria:

All consecutively hospitalized adult patients (older than 18 years of age) undergoing surgery, interventional drainage or conservative treatment, with diagnosis of cIAIs (defined as abdominal infections originating in an organ cavity, extending into the peritoneal space, and forming an abscess or peritonitis)

Exclusion Criteria:

Patients younger than 16 years-old, patients with pancreatitis or primary peritonitis

Ages: 18 Years to 110 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patients with complicated intra-abdominal infections
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2019-01-01 (Estimated); Primary Completion 2020-01-01 (Estimated); Study Completion 2020-04-01 (Estimated)

PRIMARY OUTCOMES:
Mortality rates linked to different sources of infection | 12 months
Mortality rates linked to different bacteria causing infection | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Massimo Sartelli, MD, Principal Investigator — WSES
Locations (1):
- WSES, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No